CLINICAL TRIAL: NCT06313216
Title: Efficacy of Autogenous Tooth Plates for the Treatment of Peri-implant Bone Dehiscence Following Immediate Implantation in Maxillary Esthetic Zone: Randomized Clinical Trial
Brief Title: Treatment of Peri-implant Bone Dehiscence Using Autogenous Tooth Plate
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kafrelsheikh University (Other)
Responsible Party: Principal Investigator, Walid Elamrousy, Assistant Professor of periodontology, Kafrelsheikh University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KFSIRB200-187
Record Dates: First submitted 2024-03-09; First posted 2024-03-15 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Implant Complication; Peri-Implantitis; Periodontal Diseases
MeSH Terms: conditions — Peri-Implantitis; Periodontal Diseases | interventions — Bone Plates

STUDY DESIGN:
Intervention Model Description: The present study included 63 participants, aged 20 to 45, with teeth that needed to be extracted. After Kafrelsheikh University research ethics committee approval, patients were randomized into 3 groups: group I patients underwent immediate implantation with duoteck membrane, while group II was grafted by autogenous demineralized tooth graft, but group III was grafted with autogenous demineralized tooth graft with autogenous demineralized tooth plate Clinically, pink aesthetic score (PES), midfacial mucosal alterations (MFMA), stability quotient of dental implants (SQDI) were observed at baseline, six and twelve months after implantation. Moreover, baseline, 6- and 12-months alterations of radiographic horizontal buccolingual ridge width (HBLRW), facial marginal bone level (FMBL), peri-implant Density of bone (PIDB) and peri-implant vertical bone defect depth (PIVBDD) changes were assessed using cone beam computed tomography (CBCT).
Who Masked: Participant, Outcomes Assessor
Masking Description: neither participant nor the outcome assessor know the group distribution
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Immediate Implant Placement Using duoteck membrane (Experimental): after insertion of immediate implant, the dehisced bone defect will be grafted Using duoteck membrane
  Interventions: Procedure: duoteck membrane
- Immediate Implant Placement autogenous demineralized tooth graft (Experimental): after insertion of immediate implant, the dehisced bone defect will be grafted Using autogenous demineralized tooth graft
  Interventions: Procedure: autogenous demineralized tooth graft
- Immediate Implant Placement with autogenous demineralized tooth graft and tooth plate (Experimental): after insertion of immediate implant, the dehisced bone defect will be grafted Using autogenous demineralized tooth graft and autogenous demineralized tooth plate
  Interventions: Procedure: autogenous demineralized tooth graft and plate

INTERVENTIONS:
Procedure: duoteck membrane — the dehisced bone defect will be covered with duoteck membrane
  Arms: Immediate Implant Placement Using duoteck membrane
Procedure: autogenous demineralized tooth graft — the dehisced bone defect will be covered with autogenous demineralized tooth graft
  Arms: Immediate Implant Placement autogenous demineralized tooth graft
Procedure: autogenous demineralized tooth graft and plate — the dehisced bone defect will be covered with autogenous demineralized tooth graft combined with autogenous demineralized tooth plate
  Arms: Immediate Implant Placement with autogenous demineralized tooth graft and tooth plate

SUMMARY:
The current trial aim was to evaluate clinically and radiographically the changes around dental implants inserted immediately in maxillary anterior esthetic zone using a novel combination of autogenous demineralized tooth graft. with autogenous demineralized tooth plate and compared this approach to autogenous demineralized tooth graft.

The present study included 63 patients, aged 20 to 45, with teeth that needed to be extracted. After Kafrelsheikh University research ethics committee approval, patients were randomized into 3 groups: group I patients underwent immediate implantation with Duo-Teck membrane, while group II patients underwent the same procedure, but the dehisced bone defect was grafted by autogenous demineralized tooth graft. finally group III was grafted by combination of autogenous demineralized tooth graft. with autogenous demineralized tooth plate.

DETAILED DESCRIPTION:
Patients with missing teeth face the prospect of tooth replacement either through the use of removable prostheses, fixed natural teeth-supported prostheses, or implant-supported prostheses. In many circumstances, implants are the alternative to fixed or removable prosthetic appliances.

One of the various indications of implant therapy is the replacement of periodontally hopeless teeth. The successful use of dental implants for more than 3 decades has been extensively documented for both conventional and immediate implant therapy.

The installation of implants in extraction sockets was advocated as a means to reduce the number of surgical procedures; to preserve the dimensions of the alveolar ridge; to reduce the interval between the removal of the tooth and the insertion of the implant supported restoration and furthermore, it may enhance osseointegration by taking advantage of the natural bone healing process around the implant.

A variety of regenerative techniques using combinations of bone grafts and barrier membranes have been suggested to promote bone regeneration in localized defects at implants placed into extraction sockets (Mayfield 1999). Bone substitutes were used to fill the marginal void between the implant and the bone, and barrier membranes were placed to protect the site during healing.

In the presence of fenestration or dehiscence defects, the potential for spontaneous bone formation at such defects is poor, so it is advised to use augmentation procedures for bone enhancement. Bone augmentation procedures are effective in promoting bone fill and defect resolution at implants placed in post-extraction sites, and are more successful with immediate and immediate-delayed placement than with conventional delayed placement.

The current trial aim was to evaluate clinically and radiographically the changes around dental implants inserted immediately in maxillary anterior esthetic zone using a novel combination of autogenous demineralized tooth graft. with autogenous demineralized tooth plate and compared this approach to autogenous demineralized tooth graft.

ELIGIBILITY:
Inclusion Criteria:

* above the age of 18years
* presence of non-restorable maxillary anterior tooth
* had intact socket walls following tooth extraction
* the gingival biotype was thick.

Exclusion Criteria:

* history of systemic condition
* history of using bisphosphonates or other drugs that might impact bone turnover
* a history of smoking during the previous five years,
* a history of any acute infections at the surgical site,
* teeth having root resorptions

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 63 (Actual)
Dates: Start 2024-03-15 (Actual); Primary Completion 2025-10-30 (Actual); Study Completion 2025-11-15 (Actual)

PRIMARY OUTCOMES:
Stability Quotient of dental implant (SQDI) | 12-month.
  Osstell TM was used to record the primary stability.ISQ, or Implant Stability Quotient, is a scale from 1 to 100 and is a measure of the stability of an implant. The ISQ scale has a non-linear correlation to micro mobility. With more than 1400 scientific references, investigators now know that high stability means >70 ISQ, between 60-69 is medium stability and < 60 ISQ is considered as low stability.
pink esthetic score (PES) | 12-month.
  The pink esthetic score (PES) evaluates the esthetic outcome of soft tissue around implant-supported single crowns in the anterior zone by awarding seven points for the mesial and distal papilla, soft-tissue level, soft-tissue contour, soft-tissue color, soft-tissue texture, and alveolar process deficiency.Using a 0-1-2 scoring system, 0 being the lowest, 2 being the highest value, the maximum achievable PES was 14
facial marginal bone level (FMBL) | 12-month.
  Utilizing CBCT sagittal sections, the BMBL was evaluated by computerized analysis. Navigation was done on the multiplanar display until the implant's precise same-view location was established on the reformatted cross-sectional section and panoramic view.

CONTACTS AND LOCATIONS:
Overall Officials: Walid AH Elamrousy, PhD, Principal Investigator — Faculty of Oral and Dental Medicine, Kafrelsheikh University
Locations (1):
- faculty of dentistry, kafrelsheikh University, Kafr ash Shaykh, Kafrelsheikh, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
undecided